CLINICAL TRIAL: NCT01730443
Title: Biomarkers of Injury and Outcome in ProTECT III (BIO-ProTECT)
Brief Title: Blood Biomarkers of Injury and Outcome in Traumatic Brain Injury
Acronym: BIO-ProTECT
Status: Terminated | Type: Observational
Why Stopped: Parent trial (ProTECT III) stopped for futility
Sponsor: Emory University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Michael Frankel, Professor, Emory University
Other Study IDs: IRB00014409a; 1R01NS071867 (NIH)
Record Dates: First submitted 2011-07-26; First posted 2012-11-21 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — with consent there will be long term storage of serum for Non-DNA testing
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- On progesterone treatment: The group assigned to progesterone treatment.
- group assigned to placebo: The group that will not be receiving progesterone treatment

SUMMARY:
Blood samples will be drawn on traumatic brain injury patients who are participating in the ProTECT III study.

DETAILED DESCRIPTION:
Blood samples will be drawn on traumatic brain injury patients who are participating in the ProTECT III study just prior to the initiation of the study drug infusion and 24 and 48 hours from the time they are enrolled in the study to test for biomarkers that may help predict how severe the injury is and how well they improve. The investigators will also test to see if the study medication is being absorbed and is staying at a consistent level in the blood stream.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe brain injury (iGCS 12-4 or motor response 2-5 if intubated).
* Age >18 years (or developmental stage Tanner 5 in patients where age is not known)
* Blunt, traumatic, closed head injury (altered mental status due to brain injury)
* Able to initiate study drug infusion within 4 hours from time of injury -

Exclusion Criteria:

* Non-survivable injury as determined by treating
* Bilateral dilated unresponsive pupils
* Spinal cord injury with neurological deficits, pre-injury paralysis (quad/paraplegic)
* Inability to perform activities of daily living (ADL) without assistance
* Cardiopulmonary arrest
* Status epilepticus on arrival or concern for post ictal state
* systolic blood pressure < 90 for two consecutive readings at least 5 minutes apart any time prior to randomization
* O2 Sat < 90 for at least 5 consecutive minutes any time prior to randomization
* Prisoner or ward of state
* Known active breast or reproductive organ cancers (via medical records or family interview)
* Known allergy to progesterone or Intralipid components (egg yolk) (via medical records or family interview)
* Known history of blood clotting disorder (Protein S or C deficiency, etc.) or history of pulmonary embolism (via medical records or family interview) or active/ongoing thromboembolic event (myocardial infarction, ischemic stroke, pulmonary embolism, deep vein thrombosis).
* Blood or serum ethanol (EtOH) ≥ 250 mg %
* Positive qualitative urine or serum pregnancy test
* Concern for inability to follow up at 6 months (residence in foreign country, homeless with limited contacts,
* undocumented immigrants, or high likelihood of becoming incarcerated during study period, etc.)
* Patient in Opt Out registry or wearing Opt Out bracelet -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a moderate to severe blunt traumatic brain injury who meet the inclusion and exclusion criteria for the ProTECT III study.
Sampling Method: Probability Sample
Enrollment: 576 (Actual)
Dates: Start 2011-07; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
serum biomarkers of structural brain injury (S100B, glial fibrillary acid protein, ubiquitin carboxyl-terminal esterase L1, SBDP150) and progesterone levels will be measured. | Baseline, 24 hours, 48 hours
  Blood will be collected/processed at baseline, 24 hours and 48 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Frankel, MD, Principal Investigator — Emory University
Locations (37):
- United States (37):
  - Banner Good Samaritan Health Center, Phoenix, Arizona
  - Maricopa Integrated Health System, Phoenix, Arizona
  - Scottsdale Healthcare, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - Stanford Medical Center, Palo Alto, California
  - San Francisco General Hospital, San Francisco, California
  - Regional Medical Ctr.-San Jose, San Jose, California
  - Santa Clara Valley Medical Center, San Jose, California
  - Grady Memorial Hospital, Atlanta, Georgia
  - University of Kentucky Hospital, Lexington, Kentucky
  - University of Maryland Shock Trauma, Baltimore, Maryland
  - Johns Hopkins, Baltimore, Maryland
  - Detroit Receiving, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Sinai Grace Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Beaumont Health System, Royal Oak, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Hospital, Robbinsdale, Minnesota
  - Regions Medical Center, Saint Paul, Minnesota
  - St. Johns Mercy Medical Center, St Louis, Missouri
  - NYP Columbia, New York, New York
  - University Hospital, Cincinnati, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - St. Lukes Hospital, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Jefferson Hospital, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Regional Medical Center/Elvis Presley Memorial Trauma Center, Memphis, Tennessee
  - Brackenridge Hospital, Austin, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - Brooke Army Medical Center, San Antonio, Texas
  - Virginia Commonwealth, Richmond, Virginia
  - Froederdt Memorial Hospital, Milwaukee, Wisconsin